CLINICAL TRIAL: NCT06634225
Title: IMUSEP : Use of Inertial Navigation Systems to Detect and Characterize Early Locomotor Disorders in Patients With Multiple Sclerosis.
Brief Title: Use of Inertial Units in Patient With Multiple Sclerosis (IMUSEP)
Acronym: IMUSEP
Status: Recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: RC-P00121
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Medical Device; Coordination and Balance Disturbances
Keywords: Multiple Sclerosis; Trigno Avanti Sensor; Coordination and Balance Disturbances
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Volunteers: Volunteers without pathology
  Interventions: Diagnostic Test: Usual care (as recommended by the Haute Authorité de Santé (HAS)) and medical device test
- Patient with multiple sclerosis: Patient with multiple sclerosis
  Interventions: Diagnostic Test: Usual care (as recommended by the Haute Authorité de Santé (HAS)) and medical device test

INTERVENTIONS:
Diagnostic Test: Usual care (as recommended by the Haute Authorité de Santé (HAS)) and medical device test — Patients will receive the care they need, in line with HAS recommendations. They will be asked to perform two gait analysis tests on a three-dimensional platform, equipped with sensors (medical device).
  Groups: Patient with multiple sclerosis
Diagnostic Test: Usual care (as recommended by the Haute Authorité de Santé (HAS)) and medical device test — They will be asked to perform two gait analysis tests on a three-dimensional platform, equipped with sensors (medical device).
  Groups: Volunteers

SUMMARY:
The goal of this case control study is to evaluate the use of inertial navigation systems to detect and characterize early locomotor disorders in patients with multiple sclerosis (MS). The study aims to:

• Validate the contribution and inefficiency indexes obtained by the Trigno® Avanti Sensor inertial units, in comparison with indexes calculated with 3D motion analysis during walking and tandem in early-stage MS patients.

Researchers will compare MS patients, to healthy controls.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory disease of the central nervous system, and the leading cause of non-traumatic neurological disability in young adults. It affects around 100,000 people in France, and 5,000 are newly diagnosed each year. It generally begins between the ages of 20 and 40, and mainly affects women (sex ratio 3 women/1 man).

The clinical presentation of MS is highly polymorphic. Patients may present with motor deficits, sensory disorders, spasticity, gait disorders, balance disorders, visual disturbances, etc. The symptoms that have the greatest impact on patients' quality of life in the first 5 years following diagnosis are gait and balance disorders. However, these early disorders are barely visible on clinical examination, and are not highlighted by the balance and gait tests frequently used in routine practice. These sub-clinical locomotor disorders are also not taken into account by the Expanded Disability Status Scale (EDSS). However, the discomfort reported by patients is objectified using the Multiple Sclerosis Walking Scale-12 (MSWS-12) questionnaire.

The management of balance and gait disorders is essential to limit deconditioning during exercise and reduce their impact on patients' quality of life. Detecting these disorders is therefore a key factor in improving our understanding of them, and enabling us to provide appropriate rehabilitation.

In the early stages, gait and balance disorders can be detected by means of three-dimensional movement analysis.

Certain parameters, such as contribution and inefficiency indexes, have proved useful in detecting and quantifying gait and balance disorders in early-stage MS patients. These indexes are based on the calculation of linear moments. The contribution index reflects the contribution of each body segment to body forward motion, while the inefficiency index reflects the motor performance of a segment in carrying out a locomotor task. These indices could provide physical markers for quantifying balance and gait disorders and their progression, and thus help in disease monitoring.

However, 3D motion analysis is costly in both human and technical terms, and is restricted to a laboratory environment.

At present, in France, movement analysis laboratories are not widely available for clinical evaluation, which limits the screening of balance and gait disorders in the early stages of MS, and their follow-up in private practice. On the other hand, inertial measurement systems are inexpensive, easy-to-use tools that could help detect balance and gait disorders at an early stage in MS. In fact, inertial units comprise at least an accelerometer and a gyroscope, which can also be combined with a magnetometer. The kinematics of body segments could be used to calculate contribution and inefficiency indexes, in an ecological approach geared towards everyday practice, thus democratizing and facilitating the monitoring of these disorders.

In this study, the medical device used is Trigno® Avanti Sensor. This research evaluates a medical strategy that would enable to validate the transposition of a method for calculating contribution and inefficiency indexes from data obtained by the medical device.

ELIGIBILITY:
Inclusion Criteria for patient:

* Age 18 to 65 (inclusive)
* Expanded Disability Status Scale (EDSS) ≤ 4
* Proficient in French
* Agreeing to participate in the study and having signed the informed consent form
* Affiliated with a social security scheme

Inclusion Criteria for Volunteers:

* Age 18 to 65 (inclusive)
* Proficient in French
* Agreeing to participate in the study and having signed the informed consent form
* Affiliated with a social security plan

Exclusion Criteria for patient:

* MS crisis within the last 6 weeks
* Botulinum toxin injection in the last 3 months
* Neurological pathology other than MS
* Disabling musculoskeletal pathology
* Unstable cardiac and respiratory pathology
* Pregnant women
* Patients with comprehension or cognitive disorders
* Recent change in background treatment (< 3 months)
* Patients under guardianship or curatorship
* Presence of implanted electronic devices of any kind, including pacemakers or similar assistive devices, electronic infusion pumps and implanted pacemakers
* Allergy to silver

Exclusion Criteria for Volunteers:

* Neurological pathology
* Rheumatological pathology
* Antecedent of sprains (< 3 months), fractures (< 1 year) in the lower limbs
* Pregnant women
* Person under guardianship or trusteeship
* Presence of implanted electronic devices of any kind, including pacemakers or similar assistive devices electronic infusion pumps and implanted pacemakers
* Allergy to silver

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis patients and volunteers
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-11-11 (Estimated); Study Completion 2025-11-11 (Estimated)

PRIMARY OUTCOMES:
Intra-class correlation coefficients (ICC) and their 95% confidence intervals (IC95%) for validity of the Trigno® Avanti Sensor | 1 month
  Intra-class correlation coefficients (ICC) and their 95% confidence intervals (IC95%) will be calculated to validate the contribution and inefficiency indexes obtained by the Trigno® Avanti Sensor inertial units, in comparison with indexes calculated with 3D motion analysis during walking and tandem in early-stage MS patients, and in healthy controls. The coefficient are interpreted as follows:
  (>0.8) very high correlation, (0.61-0.79) good correlation, moderate correlation, (0.41-0.60) low correlation if less bad correlation.
  These quantified indexes could be used as physical markers to quantify both the balance deterioration and the efficiency of rehabilitation program during the follow up of MS from the early stage of their disease..

SECONDARY OUTCOMES:
Intra-class correlation coefficients (ICC) and their 95% confidence intervals (IC95%) for repeatability | 1 month
  Intra-class correlation coefficients (ICC) and their 95% confidence intervals (IC95%) will be calculated to evaluate the repeatability of measures of theTrigno® Avanti Sensor inertial units comparing at baseline and at one months.
Intra-class correlation coefficients (ICC) and their 95% confidence intervals (IC95% )for the whole-body angular momentum | Baseline, 1 month
  Evaluate the agreement between whole-body angular momentum during walking and tandem walking calculated with Trigno® Avanti Sensor inertial units and 3D motion analysis in MS patients and healthy controls.
Intra-class correlation coefficients (ICC) and their 95% confidence intervals (IC95%) between the Expanded Disability Status Scale (EDSS) and the contribution and inefficiency indexes | 1 month
  Evaluate the correlation between the EDSS and the contribution and inefficiency indexes for each each method (Trigno® Avanti Sensor inertial units/3D analysis).
Intra-class correlation coefficients (ICC) and their 95% confidence intervals (IC95%) between the MSWS-12 (multiple sclerosis walking scale-two weeks) and the contribution and inefficiency indexes | 1 month
  Assess the correlation between discomfort reported by MS patients and the contribution and inefficiency indexes, for each method method (Trigno® Avanti Sensor inertial units / 3D).
Intra-class correlation coefficients (ICC) and their 95% confidence intervals (IC95%) between the MSWS-12 and whole-body angular momentum method (Trigno® Avanti Sensor inertial units / 3D 3D). | 1 month
  Evaluate the correlation between discomfort reported by MS patients and whole-body angular momentum for each method (Trigno® Avanti Sensor inertial units/3D analysis).
Differences in contribution and inefficiency indexes between groups | 1 month
  Evaluate the ability of Trigno® Avanti Sensor inertial sensors to detect the same differences between MS patients and healthy controls as 3D motion analysis.
  These quantified indexes could be used as physical markers to quantify both the balance deterioration and the efficiency of rehabilitation program during the follow up of MS from the early stage of their disease..

CONTACTS AND LOCATIONS:
Overall Officials: Caroline MASSOT, PhD, Principal Investigator — Hôpital Saint-Philibert
Locations (2):
- France (2):
  - Saint-Philibert Hospital, Lomme, Hauts-de-France
  - Saint-Amand-Les-Eaux Hospital, Saint-Amand-les-Eaux, Hauts-de-France

IPD SHARING:
Plan to Share IPD: No